CLINICAL TRIAL: NCT02940327
Title: A Feasibility Study to Consider the Relationship Between Markers of Red Cell Damage, Inflammation and the Recovery Process of Newborns Requiring Extracorporeal Membrane Oxygenation (ECMO) for Persistent Pulmonary Hypertension of the Newborn (PPHN): Mi-ECMO
Brief Title: Markers of Inflammation and Lung Recovery in ECMO Patients for PPHN
Acronym: Mi-ECMO
Status: Completed | Type: Observational
Sponsor: University of Leicester (Other)
Collaborators: University Hospitals, Leicester (Other); Heart Link Children's Charity (Other); British Heart Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 0553
Record Dates: First submitted 2016-10-13; First posted 2016-10-20 (Estimated); Results first posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2018-05

CONDITIONS: Persistent Pulmonary Hypertension of the Newborn
Keywords: ECMO; PPHN; Pulmonary Hypertension of the Newborn; Markers of inflammation; Mi-Ecmo
MeSH Terms: conditions — Persistent Fetal Circulation Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples, Urine samples, Respiratory samples
Oversight: Data Monitoring Committee: No

SUMMARY:
Respiratory failure in newborns is common and has high rates of death. Where conventional intensive care strategies have failed, newborn children are referred to treatment with Extra- Corporeal Membrane Oxygenation (ECMO). This involves connecting children via large bore cannulas placed in their heart and major blood vessels to an artificial lung that adds oxygen to their blood and removes waste gases (carbon dioxide). Although this treatment saves lives, it still has some limitations. In particular, severe complications like bleeding, or damage to the kidneys can occur. These complications can lead to death in some cases and long-term disability in others. Based on ongoing research in adults and children undergoing cardiac surgery the investigators have identified a new process that may underlie some of the complications observed in ECMO. The investigators have noted that when transfused blood is infused in an ECMO circuit, this results in the accelerated release of substances from the donor cells that cause organ damage; at least in adults. There are treatments that can reverse this process. Before the investigators explore whether these treatments should be used in newborn children on ECMO, the investigators must first demonstrate that they can measure the complex inflammatory processes that occur in these critically ill children. The investigators therefore propose to conduct a feasibility study to identify the practical issues and challenges that would need to be overcome in order to perform a successful trial in this high-risk population.

DETAILED DESCRIPTION:
The primary hypothesis is that damage to red blood cells by the exposure to the ECMO circuit will result in inflammatory responses that mitigate against successful weaning from Extra-Corporeal Membrane Oxygenation (ECMO) for Persistent Pulmonary Hypertension of the Newborn (PPHN).

The secondary hypothesis are:

1. Damage to red cells will result in platelet, leukocyte and endothelial activation.
2. Markers of platelet, endothelial and leukocyte activation are indicators of lung inflammation and injury severity and hence lung recovery.
3. Markers of platelet, endothelial and leukocyte activation are indicators of kidney injury severity and hence acute kidney injury.
4. The level of oxidative stress will correlate with type shifts in pulmonary macrophages, tissue iron deposition and organ injury.
5. Ability to raise anti-oxidative response, measured by Heme Oxigenase-1 (HMOX 1) expression, will correlate with shorter intubation times and less severe kidney and lung injury.
6. Granulocyte and platelets activation are secondary to rising redox potential and the levels of activation will correlate with longer intubation times and more severe organ injury.
7. Markers of anti-oxidative response, platelet, endothelial and leukocyte activation, as well as oxidative stress levels have diagnostic and prognostic utility for the prediction of key clinical events including delayed time to recovery, acute kidney injury in paediatric patients undergoing Extra-Corporeal Membrane Oxygenation (ECMO) for Persistent Pulmonary Hypertension of the Newborn (PPHN).

This is a pilot feasibility study that will establish the following:

1. Recruitment rates and patient flows for 24 patients specified as the target population for the feasibility study
2. Withdrawal rate, and completeness of follow-up and data collection in a paediatric population at high risk for death and major morbidity
3. The proportions (categorical data) and variance (continuous data) for the primary and secondary outcomes of interest. These will be used to model the sample sizes and outcomes that may be used in a definitive study
4. Perceptions of family members whose children participate in the study as to the appropriateness of the screening and consent process

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of PPHN
2. Patients that require ECMO support as determined by the ECMO team
3. Patients aged less than 30 days
4. Emergency consent obtained within 12 hours from cannulation, and ultimately full consent

Exclusion Criteria:

1. PPHN is caused by a congenital heart pathology
2. ECMO is required for a congenital heart disease
3. Lack of consent

Max Age: 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study will be conducted at a regional ECMO centre in the UK, the University Hospitals of Leicester NHS Trust. This unit performs over 60 neonatal and paediatric ECMO per year, of which at least 40 are expected to be performed for the treatment of PPHN in infants.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2016-02-19; Primary Completion 2017-07-10 (Actual); Study Completion 2017-07-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of Leicester NHS Trust, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
statistical analysis

REFERENCES:
- [Background] Mamikonian LS, Mamo LB, Smith PB, Koo J, Lodge AJ, Turi JL. Cardiopulmonary bypass is associated with hemolysis and acute kidney injury in neonates, infants, and children*. Pediatr Crit Care Med. 2014 Mar;15(3):e111-9. doi: 10.1097/PCC.0000000000000047. PMID 24394997
- [Background] Schaible T, Hermle D, Loersch F, Demirakca S, Reinshagen K, Varnholt V. A 20-year experience on neonatal extracorporeal membrane oxygenation in a referral center. Intensive Care Med. 2010 Jul;36(7):1229-34. doi: 10.1007/s00134-010-1886-5. Epub 2010 Apr 28. PMID 20425105
- [Background] Mugford M, Elbourne D, Field D. Extracorporeal membrane oxygenation for severe respiratory failure in newborn infants. Cochrane Database Syst Rev. 2008 Jul 16;(3):CD001340. doi: 10.1002/14651858.CD001340.pub2. PMID 18646070
- [Background] Konduri GG, Kim UO. Advances in the diagnosis and management of persistent pulmonary hypertension of the newborn. Pediatr Clin North Am. 2009 Jun;56(3):579-600, Table of Contents. doi: 10.1016/j.pcl.2009.04.004. PMID 19501693
- [Background] Bahrami KR, Van Meurs KP. ECMO for neonatal respiratory failure. Semin Perinatol. 2005 Feb;29(1):15-23. doi: 10.1053/j.semperi.2005.02.004. PMID 15921148
- [Background] UK collaborative randomised trial of neonatal extracorporeal membrane oxygenation. UK Collaborative ECMO Trail Group. Lancet. 1996 Jul 13;348(9020):75-82. PMID 8676720
- [Background] Zwiers AJ, de Wildt SN, Hop WC, Dorresteijn EM, Gischler SJ, Tibboel D, Cransberg K. Acute kidney injury is a frequent complication in critically ill neonates receiving extracorporeal membrane oxygenation: a 14-year cohort study. Crit Care. 2013 Jul 24;17(4):R151. doi: 10.1186/cc12830. PMID 23883698
- [Background] Lazar DA, Cass DL, Olutoye OO, Welty SE, Fernandes CJ, Rycus PT, Lee TC. The use of ECMO for persistent pulmonary hypertension of the newborn: a decade of experience. J Surg Res. 2012 Oct;177(2):263-7. doi: 10.1016/j.jss.2012.07.058. Epub 2012 Aug 10. PMID 22901797
- [Background] McNally H, Bennett CC, Elbourne D, Field DJ; UK Collaborative ECMO Trial Group. United Kingdom collaborative randomized trial of neonatal extracorporeal membrane oxygenation: follow-up to age 7 years. Pediatrics. 2006 May;117(5):e845-54. doi: 10.1542/peds.2005-1167. Epub 2006 Apr 24. PMID 16636114
- [Background] Farrow KN, Fliman P, Steinhorn RH. The diseases treated with ECMO: focus on PPHN. Semin Perinatol. 2005 Feb;29(1):8-14. doi: 10.1053/j.semperi.2005.02.003. PMID 15921147
- [Background] Bendapudi P, Rao GG, Greenough A. Diagnosis and management of persistent pulmonary hypertension of the newborn. Paediatr Respir Rev. 2015 Jun;16(3):157-61. doi: 10.1016/j.prrv.2015.02.001. Epub 2015 Feb 10. PMID 25765845
- [Background] Puthiyachirakkal M, Mhanna MJ. Pathophysiology, management, and outcome of persistent pulmonary hypertension of the newborn: a clinical review. Front Pediatr. 2013 Sep 2;1:23. doi: 10.3389/fped.2013.00023. PMID 24400269
- [Background] McILwain RB, Timpa JG, Kurundkar AR, Holt DW, Kelly DR, Hartman YE, Neel ML, Karnatak RK, Schelonka RL, Anantharamaiah GM, Killingsworth CR, Maheshwari A. Plasma concentrations of inflammatory cytokines rise rapidly during ECMO-related SIRS due to the release of preformed stores in the intestine. Lab Invest. 2010 Jan;90(1):128-39. doi: 10.1038/labinvest.2009.119. Epub 2009 Nov 9. PMID 19901912
- [Background] Fortenberry JD, Bhardwaj V, Niemer P, Cornish JD, Wright JA, Bland L. Neutrophil and cytokine activation with neonatal extracorporeal membrane oxygenation. J Pediatr. 1996 May;128(5 Pt 1):670-8. doi: 10.1016/s0022-3476(96)80133-8. PMID 8627440
- [Background] Mildner RJ, Taub N, Vyas JR, Killer HM, Firmin RK, Field DJ, Kotecha S. Cytokine imbalance in infants receiving extracorporeal membrane oxygenation for respiratory failure. Biol Neonate. 2005;88(4):321-7. doi: 10.1159/000087630. Epub 2005 Aug 18. PMID 16113527
- [Background] Graulich J, Walzog B, Marcinkowski M, Bauer K, Kossel H, Fuhrmann G, Buhrer C, Gaehtgens P, Versmold HT. Leukocyte and endothelial activation in a laboratory model of extracorporeal membrane oxygenation (ECMO). Pediatr Res. 2000 Nov;48(5):679-84. doi: 10.1203/00006450-200011000-00021. PMID 11044491
- [Background] Golej J, Winter P, Schoffmann G, Kahlbacher H, Stoll E, Boigner H, Trittenwein G. Impact of extracorporeal membrane oxygenation modality on cytokine release during rescue from infant hypoxia. Shock. 2003 Aug;20(2):110-5. doi: 10.1097/01.shk.0000075571.93053.2c. PMID 12865653
- [Background] Butler J, Pathi VL, Paton RD, Logan RW, MacArthur KJ, Jamieson MP, Pollock JC. Acute-phase responses to cardiopulmonary bypass in children weighing less than 10 kilograms. Ann Thorac Surg. 1996 Aug;62(2):538-42. PMID 8694619
- [Background] Kozik DJ, Tweddell JS. Characterizing the inflammatory response to cardiopulmonary bypass in children. Ann Thorac Surg. 2006 Jun;81(6):S2347-54. doi: 10.1016/j.athoracsur.2006.02.073. PMID 16731102
- [Background] Day JR, Taylor KM. The systemic inflammatory response syndrome and cardiopulmonary bypass. Int J Surg. 2005;3(2):129-40. doi: 10.1016/j.ijsu.2005.04.002. Epub 2005 Aug 1. PMID 17462274
- [Background] Warren OJ, Smith AJ, Alexiou C, Rogers PL, Jawad N, Vincent C, Darzi AW, Athanasiou T. The inflammatory response to cardiopulmonary bypass: part 1--mechanisms of pathogenesis. J Cardiothorac Vasc Anesth. 2009 Apr;23(2):223-31. doi: 10.1053/j.jvca.2008.08.007. Epub 2008 Oct 19. No abstract available. PMID 18930659
- [Background] Warren OJ, Watret AL, de Wit KL, Alexiou C, Vincent C, Darzi AW, Athanasiou T. The inflammatory response to cardiopulmonary bypass: part 2--anti-inflammatory therapeutic strategies. J Cardiothorac Vasc Anesth. 2009 Jun;23(3):384-93. doi: 10.1053/j.jvca.2008.09.007. Epub 2008 Dec 3. No abstract available. PMID 19054695
- [Background] Williams DC, Turi JL, Hornik CP, Bonadonna DK, Williford WL, Walczak RJ, Watt KM, Cheifetz IM. Circuit oxygenator contributes to extracorporeal membrane oxygenation-induced hemolysis. ASAIO J. 2015 Mar-Apr;61(2):190-5. doi: 10.1097/MAT.0000000000000173. PMID 25419829
- [Background] Omar HR, Mirsaeidi M, Socias S, Sprenker C, Caldeira C, Camporesi EM, Mangar D. Plasma Free Hemoglobin Is an Independent Predictor of Mortality among Patients on Extracorporeal Membrane Oxygenation Support. PLoS One. 2015 Apr 22;10(4):e0124034. doi: 10.1371/journal.pone.0124034. eCollection 2015. PMID 25902047
- [Background] Lou S, MacLaren G, Best D, Delzoppo C, Butt W. Hemolysis in pediatric patients receiving centrifugal-pump extracorporeal membrane oxygenation: prevalence, risk factors, and outcomes. Crit Care Med. 2014 May;42(5):1213-20. doi: 10.1097/CCM.0000000000000128. PMID 24351369
- [Background] Lubnow M, Philipp A, Foltan M, Bull Enger T, Lunz D, Bein T, Haneya A, Schmid C, Riegger G, Muller T, Lehle K. Technical complications during veno-venous extracorporeal membrane oxygenation and their relevance predicting a system-exchange--retrospective analysis of 265 cases. PLoS One. 2014 Dec 2;9(12):e112316. doi: 10.1371/journal.pone.0112316. eCollection 2014. PMID 25464516
- [Background] Maslach-Hubbard A, Bratton SL. Extracorporeal membrane oxygenation for pediatric respiratory failure: History, development and current status. World J Crit Care Med. 2013 Nov 4;2(4):29-39. doi: 10.5492/wjccm.v2.i4.29. eCollection 2013 Nov 4. PMID 24701414
- [Background] Toomasian JM, Bartlett RH. Hemolysis and ECMO pumps in the 21st Century. Perfusion. 2011 Jan;26(1):5-6. doi: 10.1177/0267659110396015. No abstract available. PMID 21177726
- [Background] Smith A, McCulloh RJ. Hemopexin and haptoglobin: allies against heme toxicity from hemoglobin not contenders. Front Physiol. 2015 Jun 30;6:187. doi: 10.3389/fphys.2015.00187. eCollection 2015. PMID 26175690
- [Background] Schaer DJ, Vinchi F, Ingoglia G, Tolosano E, Buehler PW. Haptoglobin, hemopexin, and related defense pathways-basic science, clinical perspectives, and drug development. Front Physiol. 2014 Oct 28;5:415. doi: 10.3389/fphys.2014.00415. eCollection 2014. PMID 25389409
- [Background] Hanssen SJ, van de Poll MC, Houben AJ, Windsant IC, Snoeijs MG, Bekers O, Buurman WA, Jacobs MJ. Hemolysis compromises nitric oxide-dependent vasodilatory responses in patients undergoing major cardiovascular surgery. Thorac Cardiovasc Surg. 2012 Jun;60(4):255-61. doi: 10.1055/s-0031-1299571. Epub 2012 Mar 12. PMID 22411759
- [Background] Rother RP, Bell L, Hillmen P, Gladwin MT. The clinical sequelae of intravascular hemolysis and extracellular plasma hemoglobin: a novel mechanism of human disease. JAMA. 2005 Apr 6;293(13):1653-62. doi: 10.1001/jama.293.13.1653. PMID 15811985
- [Background] Vermeulen Windsant IC, de Wit NC, Sertorio JT, van Bijnen AA, Ganushchak YM, Heijmans JH, Tanus-Santos JE, Jacobs MJ, Maessen JG, Buurman WA. Hemolysis during cardiac surgery is associated with increased intravascular nitric oxide consumption and perioperative kidney and intestinal tissue damage. Front Physiol. 2014 Sep 8;5:340. doi: 10.3389/fphys.2014.00340. eCollection 2014. PMID 25249983
- [Background] Vermeulen Windsant IC, Hanssen SJ, Buurman WA, Jacobs MJ. Cardiovascular surgery and organ damage: time to reconsider the role of hemolysis. J Thorac Cardiovasc Surg. 2011 Jul;142(1):1-11. doi: 10.1016/j.jtcvs.2011.02.012. Epub 2011 May 13. No abstract available. PMID 21570697
- [Background] Haase M, Bellomo R, Haase-Fielitz A. Novel biomarkers, oxidative stress, and the role of labile iron toxicity in cardiopulmonary bypass-associated acute kidney injury. J Am Coll Cardiol. 2010 May 11;55(19):2024-33. doi: 10.1016/j.jacc.2009.12.046. PMID 20447525
- [Background] Irwin DC, Baek JH, Hassell K, Nuss R, Eigenberger P, Lisk C, Loomis Z, Maltzahn J, Stenmark KR, Nozik-Grayck E, Buehler PW. Hemoglobin-induced lung vascular oxidation, inflammation, and remodeling contribute to the progression of hypoxic pulmonary hypertension and is attenuated in rats with repeated-dose haptoglobin administration. Free Radic Biol Med. 2015 May;82:50-62. doi: 10.1016/j.freeradbiomed.2015.01.012. Epub 2015 Feb 2. PMID 25656991
- [Background] Brittain EL, Janz DR, Austin ED, Bastarache JA, Wheeler LA, Ware LB, Hemnes AR. Elevation of plasma cell-free hemoglobin in pulmonary arterial hypertension. Chest. 2014 Dec;146(6):1478-1485. doi: 10.1378/chest.14-0809. PMID 24945582
- [Background] Buehler PW, Baek JH, Lisk C, Connor I, Sullivan T, Kominsky D, Majka S, Stenmark KR, Nozik-Grayck E, Bonaventura J, Irwin DC. Free hemoglobin induction of pulmonary vascular disease: evidence for an inflammatory mechanism. Am J Physiol Lung Cell Mol Physiol. 2012 Aug 15;303(4):L312-26. doi: 10.1152/ajplung.00074.2012. Epub 2012 Jun 22. PMID 22728465
- [Background] Murphy GJ, Verheyden V, Wozniak M, Sullo N, Dott W, Bhudia S, Bittar N, Morris T, Ring A, Tebbatt A, Kumar T. Trial protocol for a randomised controlled trial of red cell washing for the attenuation of transfusion-associated organ injury in cardiac surgery: the REDWASH trial. Open Heart. 2016 Mar 7;3(1):e000344. doi: 10.1136/openhrt-2015-000344. eCollection 2016. PMID 26977309
- [Background] Meyer AD, Gelfond JA, Wiles AA, Freishtat RJ, Rais-Bahrami K. Platelet-derived microparticles generated by neonatal extracorporeal membrane oxygenation systems. ASAIO J. 2015 Jan-Feb;61(1):37-42. doi: 10.1097/MAT.0000000000000164. PMID 25303795
- [Background] Nascimbene A, Hernandez R, George JK, Parker A, Bergeron AL, Pradhan S, Vijayan KV, Civitello A, Simpson L, Nawrot M, Lee VV, Mallidi HR, Delgado RM, Dong JF, Frazier OH. Association between cell-derived microparticles and adverse events in patients with nonpulsatile left ventricular assist devices. J Heart Lung Transplant. 2014 May;33(5):470-7. doi: 10.1016/j.healun.2014.01.004. Epub 2014 Jan 19. PMID 24656391
- [Background] Chung J, Suzuki H, Tabuchi N, Sato K, Shibamiya A, Koyama T. Identification of tissue factor and platelet-derived particles on leukocytes during cardiopulmonary bypass by flow cytometry and immunoelectron microscopy. Thromb Haemost. 2007 Aug;98(2):368-74. PMID 17721619
- [Background] Fu L, Hu XX, Lin ZB, Chang FJ, Ou ZJ, Wang ZP, Ou JS. Circulating microparticles from patients with valvular heart disease and cardiac surgery inhibit endothelium-dependent vasodilation. J Thorac Cardiovasc Surg. 2015 Sep;150(3):666-72. doi: 10.1016/j.jtcvs.2015.05.069. Epub 2015 Jun 5. PMID 26145768
- [Background] Nieuwland R, Berckmans RJ, Rotteveel-Eijkman RC, Maquelin KN, Roozendaal KJ, Jansen PG, ten Have K, Eijsman L, Hack CE, Sturk A. Cell-derived microparticles generated in patients during cardiopulmonary bypass are highly procoagulant. Circulation. 1997 Nov 18;96(10):3534-41. doi: 10.1161/01.cir.96.10.3534. PMID 9396452
- [Background] Fontaine D, Pradier O, Hacquebard M, Stefanidis C, Carpentier Y, de Canniere D, Fontaine J, Berkenboom G. Oxidative stress produced by circulating microparticles in on-pump but not in off-pump coronary surgery. Acta Cardiol. 2009 Dec;64(6):715-22. doi: 10.2143/AC.64.6.2044733. PMID 20128145
- [Background] Biro E, Sturk-Maquelin KN, Vogel GM, Meuleman DG, Smit MJ, Hack CE, Sturk A, Nieuwland R. Human cell-derived microparticles promote thrombus formation in vivo in a tissue factor-dependent manner. J Thromb Haemost. 2003 Dec;1(12):2561-8. doi: 10.1046/j.1538-7836.2003.00456.x. PMID 14738565
- [Background] Larson MC, Hillery CA, Hogg N. Circulating membrane-derived microvesicles in redox biology. Free Radic Biol Med. 2014 Aug;73:214-28. doi: 10.1016/j.freeradbiomed.2014.04.017. Epub 2014 Apr 18. PMID 24751526
- [Background] Piccin A, Murphy WG, Smith OP. Circulating microparticles: pathophysiology and clinical implications. Blood Rev. 2007 May;21(3):157-71. doi: 10.1016/j.blre.2006.09.001. Epub 2006 Nov 22. PMID 17118501
- [Background] Lovren F, Verma S. Evolving role of microparticles in the pathophysiology of endothelial dysfunction. Clin Chem. 2013 Aug;59(8):1166-74. doi: 10.1373/clinchem.2012.199711. Epub 2013 Mar 25. PMID 23529703
- [Background] Yong PJ, Koh CH, Shim WS. Endothelial microparticles: missing link in endothelial dysfunction? Eur J Prev Cardiol. 2013 Jun;20(3):496-512. doi: 10.1177/2047487312445001. Epub 2012 Apr 10. PMID 22496273
- [Background] Bhutani VK. Developing a systems approach to prevent meconium aspiration syndrome: lessons learned from multinational studies. J Perinatol. 2008 Dec;28 Suppl 3:S30-5. doi: 10.1038/jp.2008.159. PMID 19057608
- [Background] Akcan-Arikan A, Zappitelli M, Loftis LL, Washburn KK, Jefferson LS, Goldstein SL. Modified RIFLE criteria in critically ill children with acute kidney injury. Kidney Int. 2007 May;71(10):1028-35. doi: 10.1038/sj.ki.5002231. Epub 2007 Mar 28. PMID 17396113
- [Background] Howie SR. Blood sample volumes in child health research: review of safe limits. Bull World Health Organ. 2011 Jan 1;89(1):46-53. doi: 10.2471/BLT.10.080010. Epub 2010 Sep 10. PMID 21346890
- [Background] Modi N, Vohra J, Preston J, Elliott C, Van't Hoff W, Coad J, Gibson F, Partridge L, Brierley J, Larcher V, Greenough A; Working Party of the Royal College of Paediatrics and Child Health. Guidance on clinical research involving infants, children and young people: an update for researchers and research ethics committees. Arch Dis Child. 2014 Oct;99(10):887-91. doi: 10.1136/archdischild-2014-306444. Epub 2014 Jun 9. No abstract available. PMID 24914095
- [Background] Brierley J, Larcher V. Emergency research in children: options for ethical recruitment. J Med Ethics. 2011 Jul;37(7):429-32. doi: 10.1136/jme.2010.040667. Epub 2011 Feb 23. PMID 21345861
- [Background] Marc-Aurele KL, Steinman SL, Ransom KM, Finer NN, Dunn LB. Evaluation of the content and process of informed consent discussions for neonatal research. J Empir Res Hum Res Ethics. 2012 Jul;7(3):78-83. doi: 10.1525/jer.2012.7.3.78. PMID 22850145
- [Background] Joffe S, Cook EF, Cleary PD, Clark JW, Weeks JC. Quality of informed consent: a new measure of understanding among research subjects. J Natl Cancer Inst. 2001 Jan 17;93(2):139-47. doi: 10.1093/jnci/93.2.139. PMID 11208884
- [Derived] Pais P, Robinson S, Majithia-Beet G, Lotto A, Kumar T, Westrope C, Sullo N, Eagle Hemming B, Joel-David L, JnTala M, Corazzari C, Grazioli L, Smallwood D, Murphy GJ, Lai FY, Wozniak MJ. Biomarkers of Inflammation and Lung Recovery in Extracorporeal Membrane Oxygenation Patients With Persistent Pulmonary Hypertension of the Newborn: A Feasibility Study. Pediatr Crit Care Med. 2020 Apr;21(4):363-372. doi: 10.1097/PCC.0000000000002173. PMID 31725531

RESULTS

PARTICIPANT FLOW:
Groups:
- 1 - Observational Case-Controls: Observational Case-Controls.
Period: Overall Study
Arm/Group | 1 - Observational Case-Controls
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 1 - Observational Case-Controls
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 24
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Gestational age [Mean (Standard Deviation); unit: weeks] | 40.6 (2.6)
Weight at birth [Mean (Inter-Quartile Range); unit: kilograms] | 3.2 [2.9 to 3.5]

OUTCOME MEASURES:

1. Primary Outcome: CD16/41
Description: Change of markers of platelet and leukocyte activation in arterial blood and analysed by flow cytometry.
Time Frame: 12 hours after ECMO commencement
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- 7+ Days; <7 Days: on ECMO
Arm/Group | 7+ Days | <7 Days
Number analyzed (Participants) | 10 | 14
percent change | 1.90 (3.52) | 1.13 (3.03)

2. Primary Outcome: CD16/41
Description: Change of markers of platelet and leukocyte activation in arterial blood and analysed by flow cytometry.
Time Frame: 24 hours after ECMO commencement
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | 7+ Days | <7 Days
Number analyzed (Participants) | 10 | 14
percentage change | 3.11 (1.9) | 0.64 (3.26)

3. Primary Outcome: CD16/41
Description: Change of markers of platelet and leukocyte activation in arterial blood and analysed by flow cytometry.
Time Frame: 48 hours after ECMO commencement
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | 7+ Days | <7 Days
Number analyzed (Participants) | 10 | 12
percentage change | 0.73 (3.86) | 0.4 (4.3)

4. Primary Outcome: CD16/41
Description: Change of markers of platelet and leukocyte activation in arterial blood and analysed by flow cytometry.
Time Frame: 72 hours after ECMO commencement
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | 7+ Days | <7 Days
Number analyzed (Participants) | 10 | 8
percentage change | 1.55 (3.37) | 0.93 (1.99)

5. Primary Outcome: CD16/41
Description: Change of markers of platelet and leukocyte activation in arterial blood and analysed by flow cytometry.
Time Frame: 24 hours after decannulation
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | 7+ Days | <7 Days
Number analyzed (Participants) | 7 | 12
percentage change | 1.56 (2.27) | 0.6 (3.98)

6. Primary Outcome: CD14/41
Description: Change of markers of platelet and leukocyte activation in arterial blood and analysed by flow cytometry.
Time Frame: 12 hours after ECMO commencement
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | 7+ Days | <7 Days
Number analyzed (Participants) | 10 | 14
percentage change | 1.5 (3.37) | 0.84 (2.97)

7. Primary Outcome: CD14/41
Description: Change of markers of platelet and leukocyte activation in arterial blood and analysed by flow cytometry.
Time Frame: 24 hours after ECMO commencement
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | 7+ Days | <7 Days
Number analyzed (Participants) | 10 | 14
percentage change | 3.02 (2.39) | 0.38 (3.48)

8. Primary Outcome: CD14/41
Description: Change of markers of platelet and leukocyte activation in arterial blood and analysed by flow cytometry.
Time Frame: 48 hours after ECMO commencement
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | 7+ Days | <7 Days
Number analyzed (Participants) | 10 | 12
percentage change | 0.29 (4.51) | 0.27 (5.78)

9. Primary Outcome: CD14/41
Description: Change of markers of platelet and leukocyte activation in arterial blood and analysed by flow cytometry.
Time Frame: 72 hours after ECMO commencement
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | 7+ Days | <7 Days
Number analyzed (Participants) | 10 | 8
percentage change | 0.72 (4.65) | 0.59 (2.73)

10. Primary Outcome: CD14/41
Description: Change of markers of platelet and leukocyte activation in arterial blood and analysed by flow cytometry.
Time Frame: 24 hours after ECMO decannulation
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | 7+ Days | <7 Days
Number analyzed (Participants) | 7 | 12
percentage change | 1.01 (3.03) | 0.40 (4.58)

11. Primary Outcome: CD64/163
Description: Change of markers of platelet and leukocyte activation in arterial blood and analysed by flow cytometry.
Time Frame: 12 hours after ECMO commencement
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | 7+ Days | <7 Days
Number analyzed (Participants) | 10 | 14
percentage change | 8.7 (2.52) | 4.65 (2.81)

12. Primary Outcome: CD64/163
Description: Change of markers of platelet and leukocyte activation in arterial blood and analysed by flow cytometry.
Time Frame: 24 hours after ECMO commencement
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | 7+ Days | <7 Days
Number analyzed (Participants) | 10 | 14
percentage change | 7.34 (5.13) | 1.89 (5.87)

13. Primary Outcome: CD64/163
Description: Change of markers of platelet and leukocyte activation in arterial blood and analysed by flow cytometry.
Time Frame: 48 hours after ECMO commencement
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | 7+ Days | <7 Days
Number analyzed (Participants) | 10 | 12
percentage change | 3.26 (4.15) | 0.92 (2.52)

14. Primary Outcome: CD64/163
Description: Change of markers of platelet and leukocyte activation in arterial blood and analysed by flow cytometry.
Time Frame: 72 hours after ECMO commencement
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | 7+ Days | <7 Days
Number analyzed (Participants) | 10 | 8
percentage change | 3.31 (3.39) | 1.9 (3.86)

15. Primary Outcome: CD64/163
Description: Change of markers of platelet and leukocyte activation in arterial blood and analysed by flow cytometry.
Time Frame: 24 hours after decannulation
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | 7+ Days | <7 Days
Number analyzed (Participants) | 7 | 12
percentage change | 3.2 (3.55) | 2.27 (2.89)

16. Secondary Outcome: Change of Serum Haemoglobin Levels
Description: Clinical and biochemical markers of organ failure
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | 7+ Days | <7 Days
Number analyzed (Participants) | 10 | 14
g/L | 151.5 (33.0) | 145.4 (41.5)

17. Secondary Outcome: Duration on ECMO
Description: Clinical and biochemical markers of organ failure
Time Frame: > 7 days or did not survive to discharge
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | 7+ Days | <7 Days
Number analyzed (Participants) | 10 | 14
hours | 292 [186 to 360] | 80 [59 to 91]

18. Secondary Outcome: Number of Participants With Acute Kidney Injury
Description: Clinical and biochemical markers of organ failure
Time Frame: >7 days or did not survive to discharge
Measure: Number; unit: participants
Arm/Group | 7+ Days | <7 Days
Number analyzed (Participants) | 10 | 14
participants | 3 | 0

19. Secondary Outcome: Heart Injury as Determined by Serum Troponin Levels
Description: Clinical and biochemical markers of organ failure
Time Frame: 12 hours after ECMO commencement
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | 7+ Days | <7 Days
Number analyzed (Participants) | 10 | 14
ng/ml | 7.89 (1.17) | 6.96 (1.14)

20. Secondary Outcome: Allogenic Red Cell Transfusion Volume
Description: Clinical and biochemical markers of organ failure
Time Frame: 24 hours after ECMO is discontinued
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | 7+ Days | <7 Days
Number analyzed (Participants) | 10 | 14
ml | 289.6 (241.0) | 479.2 (268.2)

21. Secondary Outcome: Number of Participants Requiring Non Red Cell Transfusion
Description: Clinical and biochemical markers of organ failure
Time Frame: 24 hours after ECMO is discontinued
Measure: Count of Participants; unit: Participants
Arm/Group | 7+ Days | <7 Days
Number analyzed (Participants) | 10 | 14
Participants | 10 | 10

22. Secondary Outcome: Heart Injury as Determined by Serum Troponin Levels
Description: Clinical and biochemical markers of organ failure
Time Frame: 24 hours after ECMO commencement
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | 7+ Days | <7 Days
Number analyzed (Participants) | 10 | 14
ng/ml | 3.71 (1.54) | 3.11 (1.62)

23. Secondary Outcome: Heart Injury as Determined by Serum Troponin Levels
Description: Clinical and biochemical markers of organ failure
Time Frame: 48 hours after ECMO commencement
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | 7+ Days | <7 Days
Number analyzed (Participants) | 10 | 12
ng/ml | 2.13 (1.14) | 1.81 (1.28)

24. Secondary Outcome: Heart Injury as Determined by Serum Troponin Levels
Description: Clinical and biochemical markers of organ failure
Time Frame: 72 hours after ECMO commencement
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | 7+ Days | <7 Days
Number analyzed (Participants) | 10 | 8
ng/ml | 5.51 (2.03) | 5.88 (2.09)

25. Secondary Outcome: Heart Injury as Determined by Serum Troponin Levels
Description: Clinical and biochemical markers of organ failure
Time Frame: 24 hours after decannulation
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | 7+ Days | <7 Days
Number analyzed (Participants) | 7 | 11
ng/ml | 9.54 (1.39) | 7.44 (1.41)

26. Secondary Outcome: Change of Serum Haemoglobin Levels
Description: Clinical and biochemical markers of organ failure
Time Frame: 12 hours after ECMO commencement
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | 7+ Days | <7 Days
Number analyzed (Participants) | 10 | 14
g/L | 109.64 (20.81) | 112.07 (16.33)

27. Secondary Outcome: Change of Serum Haemoglobin Levels
Description: Clinical and biochemical markers of organ failure
Time Frame: 24 hours after ECMO commencement
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | 7+ Days | <7 Days
Number analyzed (Participants) | 10 | 14
g/L | 114.30 (11.92) | 109.43 (24.52)

28. Secondary Outcome: Change of Serum Haemoglobin Levels
Description: Clinical and biochemical markers of organ failure
Time Frame: 48 hours after ECMO commencement
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | 7+ Days | <7 Days
Number analyzed (Participants) | 9 | 12
g/L | 112.56 (9.14) | 113.08 (6.32)

29. Secondary Outcome: Change of Serum Haemoglobin Levels
Description: Clinical and biochemical markers of organ failure
Time Frame: 72 hours after ECMO commencement
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | 7+ Days | <7 Days
Number analyzed (Participants) | 10 | 9
g/L | 112.90 (7.65) | 109.89 (3.79)

30. Secondary Outcome: Change of Serum Haemoglobin Levels
Description: Clinical and biochemical markers of organ failure
Time Frame: 24 hours after decannulation
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | 7+ Days | <7 Days
Number analyzed (Participants) | 8 | 13
g/L | 109.25 (11.44) | 110.23 (12.15)

ADVERSE EVENTS:
Time Frame: Until discharge from Hospital
Arm/Group | 1 - Observational Case-Controls
All-Cause Mortality (participants affected / at risk) | 3/24
Serious Adverse Events (participants affected / at risk) | 3/24
Other Adverse Events (participants affected / at risk) | 1/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1 - Observational Case-Controls (N=24)
Fatal (Congenital, familial and genetic disorders) | 1 — Hypoplastic Lungs, Left Congenital Diaphragmatic Hernia
Fatal (Congenital, familial and genetic disorders) | 1 — Pulmonary Haemorrhage
Fatal (Congenital, familial and genetic disorders) | 1 — Acute Respiratory Failure
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 - Observational Case-Controls (N=24)
Resolved (Congenital, familial and genetic disorders) | 1 (1) — Chylothorax

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-02-27): https://cdn.clinicaltrials.gov/large-docs/27/NCT02940327/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-01): https://cdn.clinicaltrials.gov/large-docs/27/NCT02940327/SAP_001.pdf